CLINICAL TRIAL: NCT01385800
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate Three Doses of ToleroMune Grass in Grass Allergic Subjects Following Challenge With Grass Allergen in an Environmental Exposure Unit
Brief Title: ToleroMune Grass Exposure Unit Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Pharm-Olam International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG002
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Grass Allergy; Rhinoconjunctivitis
Keywords: Grass allergy; Rhinoconjunctivitis; Environmental Exposure Unit; Immunotherapy; ToleroMune Grass

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Intradermal injection, 1 x 8 administrations 2 weeks apart
  Interventions: Biological: Placebo
- ToleroMune Grass Dose 1 (Experimental): Intradermal injection 1 x 8 administrations 2 weeks apart
  Interventions: Biological: ToleroMune Grass
- ToleroMune Grass Dose 2 (Experimental): Intradermal injection 1 x 8 administrations 2 weeks apart
  Interventions: Biological: ToleroMune Grass
- ToleroMune Grass Dose 3 (Experimental): Intradermal injection 1 x 8 administrations 2 weeks apart
  Interventions: Biological: ToleroMune Grass

INTERVENTIONS:
Biological: ToleroMune Grass — Intradermal injection 1 x 8 administrations 2 weeks apart
  Arms: ToleroMune Grass Dose 1; ToleroMune Grass Dose 2; ToleroMune Grass Dose 3
Biological: Placebo — Intradermal injection 1 x 8 administrations 2 weeks apart
  Arms: Placebo

SUMMARY:
Grass pollen allergens are recognised as a major cause of allergic diseases in humans and animals. Worldwide, at least 40% of allergic patients are sensitised to grass pollen allergens and between 50-90% of hayfever or seasonal allergy sufferers are allergic to grass pollen. ToleroMune Grass is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of grass allergy.

This study will look at the efficacy, safety and tolerability of three doses of ToleroMune Grass in grass allergic subjects following challenge with with grass in an Environmental Exposure Unit (EEU).

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability of ToleroMune Grass in grass allergic subjects with allergic rhinoconjunctivitis. The efficacy of ToleroMune Grass will be explored in subjects using an EEU (Environmental Exposure Unit).

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 16 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of 4 visits to the EEU at least 3 days before randomisation.

In Period 2, subjects in each cohort complying with the inclusion/exclusion criteria will be randomised to one of four groups and will receive treatment every 2 weeks (±2 days) for 14 weeks.

In Period 3, Post Treatment Challenge will consist of 4 visits to the EEU about 25 weeks after the first administration in the treatment period and assessments will be performed identical to those at the baseline challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion criteria

* Male or female, aged 18-65 years.
* Minimum 2-year documented history of rhinoconjunctivitis on exposure to grass.
* Positive skin prick test to grass allergen.
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion criteria

* History of asthma.
* A history of anaphylaxis to grassallergen.
* Subjects with an FEV1 <80% of predicted.
* Subjects who cannot tolerate baseline challenge in the EEU.
* Subjects for whom administration of epinephrine is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* A history of severe drug allergy, severe angioedema or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | Upto 25 weeks

SECONDARY OUTCOMES:
Symptom scores for nasal and non nasal symptoms | Upto 25 weeks
Skin prick testing | Upto 25 weeks
Peak Nasal Inspiratory Flow | Up to 25 weeks
Grass specific IgA | Upto 26 weeks
Grass specific IgE | Upto 26 weeks
Grass specific IgG4 | Up to 26 weeks
Adverse Events | Up tp 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD MSC FRCPC, Principal Investigator — Queen's University, Kingston, Ontario
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada